CLINICAL TRIAL: NCT03734900
Title: Comparison of Effectiveness Between Platelet Lysate and Platelet-rich Plasma on Knee Osteoarthritis: a Prospective, Randomized, Placebo-controlled Trial
Brief Title: Comparison of Effectiveness Between PL and PRP on Knee Osteoarthritis: a Prospective,Randomized,Placebo-controlled Trial
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 201803124RIPD
Record Dates: First submitted 2018-10-25; First posted 2018-11-08 (Actual); Last update posted 2021-09-20 (Actual); Status verified 2021-07

CONDITIONS: Osteoarthritis (OA) of the Knee
MeSH Terms: conditions — Osteoarthritis | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Saline injection (Placebo Comparator): Sodium Chloride injection into the study knee joint every 4 weeks for a total of 3 injections
  Interventions: Other: Saline injection
- PRP injection (Experimental): PRP injection into the study knee joint every 4 weeks for a total of 3 injections
  Interventions: Biological: PRP injection
- PL injection (Experimental): PL injection into the study knee joint every 4 weeks for a total of 3 injections Platelet lysate is the product of nature activation from autologous platelet.
  Interventions: Biological: PL injection

INTERVENTIONS:
Other: Saline injection — 5ml Placebo infusion of 0.9% Sodium Chloride
  Arms: Saline injection
Biological: PRP injection — Device: "Aeon" Acti-PRP
  5ml autologous platelet rich plasma injection
  Arms: PRP injection
Biological: PL injection — Device: "Aeon" Acti-PRP
  5ml autologous platelet lysate injection
  Arms: PL injection

SUMMARY:
This study will focus on grade I to III knee osteoarthritis by randomized controlled trials which comparing the effectiveness between placebo, autologous platelet rich plasma and autologous platelet lysate injections.

DETAILED DESCRIPTION:
The current methods for treating knee osteoarthritis include delaying the disease progression and joint replacement surgery. The usual treatment methods are mostly temporary, such as taking drug and hyaluronic acid injection. Therefore, finding the safe and effective methods will greatly reduce medical resource, medical expenses and surgery cost, etc., and restore the patient's quality of life. Platelet lysate is the product of complete activation from autologous platelet. It contains rich growth factors and cytokines such as PDGF, TGF-β, VEGF, EGF and IGF, etc. It can support cell growth and doesn't have any white blood cells in it. It is superior to the platelet rich plasma because of reducing the overall inflammatory response and pain of the patient during treatment.

ELIGIBILITY:
Inclusion Criteria:

* 50 to 80 years old
* Study Subjects must be willing to sign Informed Consent to participate in the study
* In the past month, at least seven consecutive days in the squat, standing, walking or going up and down the stairs, the most serious degree of visual analogy of the knee pain (Visual Analogue Scale) is greater than or equal to 40 (the most pain is 100, not painful is 0)
* Morning joint stiffness is less than 30 minutes
* X-ray：Grade 1-3 radiographic OA as defined by the K-L classification

Exclusion Criteria:

* Knee instability
* The knee joint is obviously deformed (> 5 degree valgus or varus deviation on X-ray)
* Clinical diagnosed as Pes tendinitis, Chondromalacia
* Taking NSAIDs or steroids (including oral and injection) within one week
* Using anticoagulant drugs for a long time
* Platelet count is less than 150,000 / UL, or coagulation disorders, prothrombin time (PT value) is less than 11 seconds or greater than 16 seconds
* Leukemia, sepsis, platelet dysfunction or other blood related diseases
* tumors, infections or the trauma before the same site
* Pregnancy

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2018-05-15 (Actual); Primary Completion 2022-05-14 (Estimated); Study Completion 2022-05-14 (Estimated)

PRIMARY OUTCOMES:
Pain score of the patient | up to 24 weeks after surgery
  Using Visual Analog Score (from 0 to 10, 0 indicate no pain and 10 indicate maximal pain) to evaluate pain of surgical wound of the patient

SECONDARY OUTCOMES:
Knee functional score | up to 24 weeks after surgery
  Using Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC)
X-ray | up to 24 weeks after surgery
  Knee X-ray image
Ultrasonic image | up to 24 weeks after surgery
  Ultrasonic-between thickness of the medial and lateral sides of the femoral condyle
adverse events | up to 24 weeks after surgery
  adverse events in clinical trial

CONTACTS AND LOCATIONS:
Overall Officials: Wu Chueh-Hung, MD, CIPS, Study Director — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan